CLINICAL TRIAL: NCT01450982
Title: A Study to Investigate the Effects of JNJ-38518168 on Methotrexate Pharmacokinetics in Rheumatoid Arthritis Participants on a Stable Methotrexate Dose
Brief Title: A Study to Investigate How JNJ-38518168 May Affect the Plasma Levels of Methotrexate in Rheumatoid Arthritis Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR018655; 38518168ARA1001 (Other: Johnson & Johnson Pharmaceutical Research & Development, L.L.C.)
Record Dates: First submitted 2011-06-13; First posted 2011-10-13 (Estimated); Last update posted 2013-05-06 (Estimated); Status verified 2013-05

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; JNJ-38518168; Methotrexate
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 001 (Experimental): JNJ-38518168 / MTX Day 1: MTX: Route=oral use single dose of participant's weekly MTX dose Days 2-15: MTX: Route=oral use single dose of participant's weekly MTX dose and of JNJ-38518168 Type=exact unit=mg number=100 form=capsule route=oral use administered daily.
  Interventions: Drug: JNJ-38518168 / MTX

INTERVENTIONS:
Drug: JNJ-38518168 / MTX — Day 1: MTX: Route=oral use, single dose of participant's weekly MTX dose

SUMMARY:
The purpose of this study is to evaluate the effects of JNJ-38518168 on the pharmacokinetics (how the body handles a drug) of methotrexate in participants with rheumatoid arthritis.

DETAILED DESCRIPTION:
This is an open-label (physician and participant will know the name of the assigned drug), multi-center, non-randomized, drug/drug interaction study of JNJ-38518168 in participants with rheumatoid arthritis (RA) on a stable oral methotrexate (MTX) dose (7.5-25 mg). The treatment phase will last 16 days. Participants will be housed in the clinic for dosing and study procedures from Day -1 to Day 2 and again from Day 14 to Day 16. Participants completing treatment will have a follow-up visit between Days 22 and 25. Participants who discontinue the study prematurely will complete the Day 22 to 25 follow-up procedures at the time of discontinuation or as soon as possible thereafter. The duration of participation in the study for an individual participant will be up to 7 weeks (including screening). Participant safety will be monitored. Day 1: A single oral dose of the participant's weekly methotrexate dose. Days 2-15: Weekly MTX co-administered with two 50-mg capsules of JNJ-38518168, administered daily.

ELIGIBILITY:
Inclusion Criteria:

* Have a body mass index (BMI) between 18 and 38 kg/m2 inclusive, and a body weight between 50-110 kg, inclusive
* Have a diagnosis of Rheumatoid Arthritis functional class I-III for at least 3 months prior to Screening
* Have been treated with and tolerated oral MTX treatment for a minimum of 3 months prior to screening and must have been on a once-weekly stable MTX dose (taken as a single dose) (between 7.5-25 mg/week) for a minimum of 1 month
* Participants may continue on stable non-steroid anti-inflammatory drugs and corticosteroid background therapy for RA or stable therapies for other conditions as prescribed by physician, provided that the doses of such therapy are stable for at least 1 month prior to screening and will remain unchanged for the entire study duration.

Exclusion Criteria:

* Have current signs or symptoms of liver or renal insufficiency or cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, psychiatric, or metabolic disturbances that are severe, progressive or uncontrolled in the study doctor's opinion
* Have been treated with a monoclonal antibody for RA or have had a serious infection with 2 weeks of the study treatment period.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-06; Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Blood levels of methotrexate | Up to approximately 7 weeks
  To assess the effect of multiple doses of JNJ-38518168 on blood levels of methotrexate

SECONDARY OUTCOMES:
Blood levels of JNJ-38518168 | Up to approximately 7 weeks
  To assess the effect of methotrexate on the blood levels of JNJ-38518168
The number of participants with adverse events | Up to approximately 7 weeks
Clinical laboratory tests | Up to approximately 7 weeks
  Blood and urine tests
Electrocardiograms | Up to approximately 7 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (4):
- United States (4):
  - Anniston, Alabama
  - Daytona Beach, Florida
  - Duncansville, Pennsylvania
  - Dallas, Texas